CLINICAL TRIAL: NCT05137288
Title: Intrathecal Atropine Versus Preoperative Intravenous Ondasetron for Prevention of Postoperative Nausea and Vomiting Due to Intrathecal Morphine in Perineal Surgery
Brief Title: Intrathecal Atropine Versus Intravenous Ondasetron in Post Operative Nausea Due to Intrathecal Morphine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shehab Mahmoud Mohamed, resident doctor at anesthesia and ICU department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00013006
Record Dates: First submitted 2021-10-13; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Perineal Surgery
MeSH Terms: interventions — Ondansetron; Atropine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients receiving intrathecal atropine (Active Comparator): Patient received intrathecal hyperbaric bupivacaine ( 10 mg ) ( 2 ml 0.5% ) with morphine 250mic and atropine sulphate 100 micwith total volume = 2.5 ml .
  Interventions: Drug: Ondansetron , atropine and bupivacaine
- patients receiving preoperative intravenous ondasetron (Active Comparator): Patient received intrathecal hyperbaric bupivacaine ( 10 mg ) ( 2 ml 0.5% with 0.5 ml normal saline with morphine 250 mic ) with total volume = 2.5 ml with giving 4 mg IV ondansetron before anesthesia ( patients with body weight more than 80 Kg may need additional 4 mg IV ) .
  Interventions: Drug: Ondansetron , atropine and bupivacaine

INTERVENTIONS:
Drug: Ondansetron , atropine and bupivacaine — Patient received intrathecal hyperbaric bupivacaine ( 10 mg ) ( 2 ml 0.5% ) with morphine 250mic and atropine sulphate 100 micwith total volume = 2.5 ml .
  Patient received intrathecal hyperbaric bupivacaine ( 10 mg ) ( 2 ml 0.5% with 0.5 ml normal saline with morphine 250 mic ) with total volume = 2.5 ml with giving 4 mg IV ondansetron before anesthesia ( patients with body weight more than 80 Kg may need additional 4 mg IV ) .

SUMMARY:
To compare between intrathecal atropine versus preoperative administration of IV ondansetron in decreasing incidence of post operative nausea and vomiting related to intrathecal opioids in post operative period in perineal surgery as regard : efficacy and side effects .

ELIGIBILITY:
Inclusion Criteria:

* Age between ( 18 - 45 ) years.
* Body mass index between ( 18.5 - 35 )
* patients undergoing perineal surgery as anal fissure , piles and rectocele
* patients receiving bupivacaine ( 20 mg / 4 ml ) as spinal anesthesia
* Patinets with physical status 1 or 2 according to ASA classification

Exclusion Criteria:

* Patient refusal .
* Any contraindication of neuraxial block as : coagulopathy , skin infection at injection site or bacteremia , hypovolemia and shock , history of allergy to L.A , sever aortic stenosis or mitral stenosis ……… etc
* Patients with physical status other than 1 and 2 according to ASA classification
* Those with history of nausea and vomiting , also those who received anti emetic drugs in last 2 hours of operation .
* Allergy to any of the drug included in this study .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
frequency of attacks of postoperative nausea and vomiting | 6-9 months
  Intrathecal atropine versus preoperative intravenous ondasetron for prevention of postoperative nausea and vomiting due to intrathecal morphine

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gybels J, Erdine S, Maeyaert J, Meyerson B, Winkelmuller W, Augustinsson L, Bonezzi C, Brasseur L, DeJongste M, Kupers R, Marchettini P, Muller-Schwefe G, Nitescu P, Plaghki L, Reig E, Spincemaille G, Thomson S, Tronnier V, Van Buyten JP. Neuromodulation of pain. A consensus statement prepared in Brussels 16-18 January 1998 by the following task force of the European Federation of IASP Chapters (EFIC). Eur J Pain. 1998;2(3):203-9. doi: 10.1016/s1090-3801(98)90016-7. No abstract available. PMID 15102380
- [Background] Baciarello M, Cornini A, Zasa M, Pedrona P, Scrofani G, Venuti FS, Fanelli G. Intrathecal atropine to prevent postoperative nausea and vomiting after Cesarean section: a randomized, controlled trial. Minerva Anestesiol. 2011 Aug;77(8):781-8. PMID 21730925